CLINICAL TRIAL: NCT02794298
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on GABA Concentration and Brain Functional Connectivity in Young Adults.
Brief Title: tDCS Effects on GABA Concentration and Brain Functional Connectivity in Young Adults
Acronym: TRAINSTIM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Physikalisch-Technische Bundesanstalt Institut Berlin (PTB) (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TRAINSTIM1.C
Record Dates: First submitted 2016-04-05; First posted 2016-06-09 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Young Adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Anodal tDCS (Experimental): Anodal stimulation during resting state fMRI
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Cathodal tDCS (Experimental): Cathodal stimulation during resting state fMRI
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- sham tDCS (Sham Comparator): Sham stimulation during resting state fMRI
  Interventions: Device: sham-tDCS

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS)
  Arms: Anodal tDCS; Cathodal tDCS
Device: sham-tDCS
  Arms: sham tDCS

SUMMARY:
The aim of this study is to investigate whether anodal tDCS over the left M1 leads to a decrease of GABA concentration and alterations of functional brain connectivity in younger people, compared to sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* unobtrusive neuropsychological screening
* age: young adults: 18-30 years

Exclusion Criteria:

* Mild cognitive impairment (MCI) or other neurological diseases
* History of severe alcoholism or use of drugs
* Severe psychiatric disorders such as depression, psychosis (if not in remission) and severe untreated medical problems
* Contraindication for MRI (claustrophobia, metallic implants, ferromagnetic metals in the body, disorders of thermoregulation, pregnant women)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement of GABA concentration by magnetic resonance spectroscopy (MRS) after anodal tDCS adjusted for baseline levels. | assessed immediately before and after a 15-min stimulation time
  Investigation whether anodal tDCS leads to a significant reduction of M1-GABA concentration in younger adults compared to sham stimulation.

SECONDARY OUTCOMES:
GABA concentration assessed by MRS after cathodal tDCS adjusted for baseline levels | assessed immediately before and after a 15-min stimulation time
  To assess stimulation effects on GABA concentration by magnetic resonance spectroscopy are measured before and after cathodal tDCS.
Resting-state functional connectivity changes | assessed during a 15-min stimulation time
  Functional connectivity as measured by resting-state fMRI during tDCS compared to sham
Genotyping of learning related polymorphisms. | assessed during baseline screening
  To assess predictors of positive reaction to brain stimulation, genotyping of several learning related polymorphisms will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Bachtiar V, Near J, Johansen-Berg H, Stagg CJ. Modulation of GABA and resting state functional connectivity by transcranial direct current stimulation. Elife. 2015 Sep 18;4:e08789. doi: 10.7554/eLife.08789. PMID 26381352
- [Background] Amadi U, Allman C, Johansen-Berg H, Stagg CJ. The Homeostatic Interaction Between Anodal Transcranial Direct Current Stimulation and Motor Learning in Humans is Related to GABAA Activity. Brain Stimul. 2015 Sep-Oct;8(5):898-905. doi: 10.1016/j.brs.2015.04.010. Epub 2015 May 1. PMID 26279408
- [Background] Stagg CJ, Bachtiar V, Amadi U, Gudberg CA, Ilie AS, Sampaio-Baptista C, O'Shea J, Woolrich M, Smith SM, Filippini N, Near J, Johansen-Berg H. Local GABA concentration is related to network-level resting functional connectivity. Elife. 2014 Mar 25;3:e01465. doi: 10.7554/eLife.01465. PMID 24668166